CLINICAL TRIAL: NCT05049733
Title: The Pharmacokinetics and Pharmacodynamics of a Single Acute Dose of a Hemp-derived Oral Product With a 1:1 Ratio of CBD:CBD-A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Cultivate Biologics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00290381
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind (Participant, Outcomes Assessor), placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Participants will start with ingestion of soft gel tablets high in CBD and CBD-A, but low in THC and THC-A. The total amount of cannabinoids ingested will be 1 mg/kg and then switch to other doses after washout periods.
  Interventions: Drug: CBD 1mg/Kg; Drug: CBD 2mg/Kg; Drug: CBD 4mg/Kg; Drug: Placebo CBD
- Arm 2 (Experimental): Participants will start with ingestion of soft gel tablets high in CBD and CBD-A, but low in THC and THC-A. The total amount of cannabinoids ingested will be 2 mg/kg and then switch to other doses after washout periods.
  Interventions: Drug: CBD 1mg/Kg; Drug: CBD 2mg/Kg; Drug: CBD 4mg/Kg; Drug: Placebo CBD
- Arm 3 (Experimental): Participants will start with ingestion of soft gel tablets high in CBD and CBD-A, but low in THC and THC-A. The total amount of cannabinoids ingested will be 4 mg/kg and then switch to other doses after washout periods.
  Interventions: Drug: CBD 1mg/Kg; Drug: CBD 2mg/Kg; Drug: CBD 4mg/Kg; Drug: Placebo CBD
- Arm 4 (Placebo Comparator): Participants will begin with ingestion of placebo soft gel tablets that do not contain cannabinoids and then switch to other doses after washout periods.
  Interventions: Drug: CBD 1mg/Kg; Drug: CBD 2mg/Kg; Drug: CBD 4mg/Kg; Drug: Placebo CBD

INTERVENTIONS:
Drug: CBD 1mg/Kg — Participants will ingest soft gel tablets containing CBD 1mg/Kg
Drug: CBD 2mg/Kg — Participants will ingest soft gel tablets containing CBD 2mg/Kg
Drug: CBD 4mg/Kg — Participants will ingest soft gel tablets containing CBD 4mg/Kg
Drug: Placebo CBD — Participants will ingest soft gel tablets containing placebo for CBD

SUMMARY:
The purpose of this study is to examine the pharmacokinetics and pharmacodynamics of a hemp-derived oral product containing cannabidiol (CBD) and cannabidiolic acid (CBD-A) at a 1:1 ratio.

DETAILED DESCRIPTION:
The purpose of the present study is to examine the pharmacokinetics and pharmacodynamics of a novel hemp-derived oral cannabinoid product, at various doses, in healthy adults. The study will utilize a within-subjects, placebo-controlled, double-blind, ascending-dose design. Drug administration will be double blind (the participant and research staff will be unaware of the dose administered). Upon enrollment, participants will complete 4 dosing conditions (placebo, 1 mg/kg, 2 mg/kg, 4 mg/kg of cannabinoids). Each condition will consist of a single acute drug exposure, followed by an 8-hour period to evaluate acute pharmacodynamic and pharmacokinetic (PK) drug effects. Biological specimens (blood and urine) will be obtained throughout these 8 hours to characterize the pharmacokinetics of CBD, CBD-A, delta-9-Tetrahydrocannabinol (THC), and THC-A, as well as other relevant cannabinoids and metabolites. Pharmacodynamic assessments including subjective drug effects, cognitive performance testing, and vital signs will also be collected for 8 hours post-drug administration. For each of the two days after each experimental session, participants will be asked to return to the lab for brief visits (~20 min) to provide additional biospecimens (~24 and ~48 hrs after dosing) to allow for further PK analysis. These procedures will be completed 4 separate times by each participant (sessions will be separated by at least 1 week to allow for sufficient drug washout between doses).

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 55
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit and again upon admission for each experimental session
5. Test negative for other drugs of abuse, including alcohol, at the screening visit and upon arrival for the experimental session
6. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission
7. Weigh between 110 lbs (50 kg) and 220 lbs (100 kg)
8. Blood pressure at screening visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
9. Self-report prior experience using cannabis or CBD products, but no cannabis, cannabinoid, or hemp product use in the prior 30 days
10. Have not donated blood in the prior 30 days
11. For women of children bearing potential and men with female partners of child-bearing potential, must be willing to use an effective form of contraception during the study and for at least 30 days after the last drug administration session

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine in the past 30 days
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures
3. Use of an over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days (or 5 half-lives for that specific drug) of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study results or the safety of the participant
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days (or 5 half-lives for that specific drug) of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the participant. This includes any medication metabolized via CYP2D6, CYP2C9, CYP2B10, or which induce/inhibit CYP3A4 enzymes.
5. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina)
6. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing
7. Epilepsy or a history of seizures.
8. Individuals with anemia for whom, in the opinion of the study team, participation would pose increased medical risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - maximum concentration (CMax) for CBD | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentration (Cmax) is determined as the highest concentration (in nanogram per milliliter, ng/mL) reached for each individual.
Pharmacokinetics - maximum concentration (CMax) for CBD-A | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentration (Cmax) is determined as the highest concentration (in nanogram per milliliter, ng/mL) reached for each individual.
Pharmacokinetics - maximum concentration (CMax) for THC | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentration (Cmax) is determined as the highest concentration (in nanogram per milliliter, ng/mL) reached for each individual.
Pharmacokinetics - maximum concentration (CMax) for THC-A | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentration (Cmax) is determined as the highest concentration (in nanogram per milliliter, ng/mL) reached for each individual.
Pharmacokinetics - AUC for CBD | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
Pharmacokinetics - AUC for CBD-A | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
Pharmacokinetics - AUC for THC | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
Pharmacokinetics - AUC for THC-A | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
Pharmacokinetics - Tmax for CBD | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The Tmax, or time to reach maximum concentration, is the timepoint at which the Cmax is observed.
Pharmacokinetics - Tmax for CBD-A | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The Tmax, or time to reach maximum concentration, is the timepoint at which the Cmax is observed.
Pharmacokinetics - Tmax for THC | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The Tmax, or time to reach maximum concentration, is the timepoint at which the Cmax is observed.
Pharmacokinetics - Tmax for THC-A | 48 hrs
  Blood cannabinoid concentrations will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The Tmax, or time to reach maximum concentration, is the timepoint at which the Cmax is observed.

SECONDARY OUTCOMES:
Driving Under the Influence of Drugs (DRUID) application global impairment score | 8 hrs
  Acute cognitive and behavioral impairment will be assessed with global impairment score(range 0-100) on the DRUID app (higher scores indicate greater impairment).
Number of Correct Trials on Paced Auditory Serial Addition Task (PASAT) | 8 hrs
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Will report the total correct trials out of 90 recorded (lower scores indicate worse performance).
Number of Correct Trials on the Digit Symbol Substitution Task (DSST) | 8 hrs
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Will report the total correct trials in 90 seconds (lower scores indicate worse performance).
Distance from Central Stimulus on the Divided Attention Task (DAT) | 8 hrs
  Computerized version of Divided Attention Task will be administered to assess divided attention. Will report the mean total distance from the central stimulus (in computer pixels) over the course of the task (higher scores indicate worse performance). Note that there is no defined upper limit to these scores.
Feel Drug Effect as assessed by the Drug Effect Questionnaire (DEQ) | 8 hrs
  The DEQ will be used to obtain subjective ratings of "feel drug effects". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No